CLINICAL TRIAL: NCT06911879
Title: The Effect of Ketogenic-Caloric Restricted Dietary Intervention on Metabolic Endotoxemia Among Prediabetic Obese Jordanian Adults Aged 18-40 Years Old: A Randomized Clinical Trial
Brief Title: The Effect of Ketogenic-caloric Restricted Diet on Metabolic Endotoxemia in Prediabetic Obese Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Aseel Basem jawamis, Principal Investigator, PhD Candidate in Human Nutrition and Dietetics, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 381/2025
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Insulin Resistance; Metabolic Endotoxemia; Inflammation Biomarkers; Ketogenic Diet; Caloric Restriction; Obesity; Prediabetes
Keywords: ketogenic diet; Ketogenic-Caloric Restricted Diet; metabolic endotoxemia; insulin resistance; obesity; prediabetes; inflammation
MeSH Terms: conditions — Insulin Resistance; Obesity; Prediabetic State; Inflammation | interventions — Diet, Ketogenic; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketogenic diet with caloric restriction (Experimental)
  Interventions: Other: Ketogenic diet with caloric restriction
- Normal diet with caloric restriction (Active Comparator)
  Interventions: Other: Normal diet with caloric restriction
- Normal diet without caloric restriction (Active Comparator)
  Interventions: Other: Normal diet without caloric restriction

INTERVENTIONS:
Other: Ketogenic diet with caloric restriction — Participants in this group will follow a ketogenic diet with caloric restriction (-550 kcal/day), consisting of approximately 5-10% carbohydrates, 15-25% protein, 70-80% fat. The daily carbohydrate intake will be limited to less than 50g per day. The intervention will last for 12 weeks, with regular dietary monitoring and adherence checks every two weeks.
  Arms: Ketogenic diet with caloric restriction
Other: Normal diet with caloric restriction — Participants in this group will follow a normal diet with caloric restriction (-550 kcal/day), consisting of approximately 45-60% carbohydrates, 15-25% protein, 20-30% fat. The intervention will last for 12 weeks, with regular dietary monitoring and adherence checks every two weeks.
  Arms: Normal diet with caloric restriction
Other: Normal diet without caloric restriction — Participants in this group will follow a normal diet without caloric restriction, consisting of approximately 45-60% carbohydrates, 15-25% protein, 20-30% fat. The intervention will last for 12 weeks, with regular dietary monitoring and adherence checks every two weeks.
  Arms: Normal diet without caloric restriction

SUMMARY:
Insulin resistance increases the risk of type 2 diabetes and cardiovascular disease, with gut dysbiosis emerging as a contributing factor. Metabolic endotoxemia, characterized by elevated serum lipopolysaccharides (LPS), disrupts insulin signaling via inflammatory pathways. While dietary interventions may lower LPS levels and improve insulin resistance, evidence on the effectiveness of ketogenic diet in this context remains limited.

This randomized controlled trial aims to assess the effects of a ketogenic-caloric restricted diet on metabolic endotoxemia, measured by serum LPS levels, in prediabetic obese Jordanian adults aged 18-40 years in Amman over 12 weeks. Ninety participants will be randomly assigned to one of three groups (n=30 each): a ketogenic-caloric restricted diet, a normal-fat caloric restricted diet, or a control group (normal-fat without caloric restriction). Anthropometric parameters and dietary intake will be evaluated at baseline, week 6, and week 12. Blood samples will be collected at baseline and week 12 for measuring fasting glucose, insulin, LPS, inflammatory cytokines. Dietary adherence will be monitored through food records. This study aims to provide new insights into the role of dietary interventions in modifying metabolic endotoxemia and improving insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females individuals aged 18-40 years

  * Individuals with a body mass index (BMI) greater than 30 kg/m² and less than 40 kg/m².
  * Individuals medically diagnosed with prediabetes by a physician prior to enrollment in the study as indicated by hemoglobin A1c (HbA1c) levels between 5.7% and 6.4% (American Diabetes Association, 2024), or HOMA-IR score of greater than 1.8.
  * Individuals demonstrating a willingness to follow the dietary protocol
  * Individuals engaging in sedentary physical activity levels

Exclusion Criteria:

* Individuals diagnosed with any other chronic disease or type 1 and type 2 diabetes mellitus.

  * Individuals have experienced weight loss of more than 5% in the last three months.
  * Pregnant or lactating women.
  * Individuals undergoing any form of drug treatment.
  * Individuals with a history of major surgery.
  * Individuals have consumed pro-/pre/symbiotic or antibiotics in the past three months.
  * Individuals who engage in any form of regular sports activity.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Serum Lipopolysaccharides (LPS) Levels | Baseline and after 12 weeks of intervention
  Serum LPS levels will be measured using ELISA before and after the dietary intervention to assess the impact of ketogenic-caloric restricted diet on metabolic endotoxemia in adult participants with obesity and insulin resistance."

SECONDARY OUTCOMES:
TNF-α, IL-6 serum levels | Baseline and after 12 weeks of intervention
  Serum TNF-α and IL-6 levels will be measured using ELISA at baseline and after 12 weeks to assess the inflammatory response to dietary interventions.
Change in Fasting Glucose Level | Baseline and after 12 weeks of intervention
  Fasting glucose will be measured to assess glycemic control before and after the dietary intervention.
Lipid Profile (Total Cholesterol, LDL, HDL, Triglycerides) | Baseline and after 12 weeks of intervention
  Lipid profile, including total cholesterol, LDL, HDL, and triglycerides, will be analyzed at baseline and post-intervention to determine the impact of dietary modifications on lipid metabolism.
Ketone bodies | week 6 and after 12 weeks of intervention
  ketone bodies will be measured to assess the adherence to ketogenic diet (just for arm 1) levels at week 6 and after 12 weeks of intervention."
Change in Body weight in kilograms | Baseline and every 2 weeks until week 12
  Body weight in kilograms will be measured using a calibrated digital scale (InBody 120) while participants are wearing light clothing and no shoes. Measurements will be taken every two weeks throughout the 12-week intervention period.
  The average weight will be recorded at each time point, and changes from baseline will be analyzed across intervention groups.
Dietary Intake using Food Records | week4, week 8 and week 12
Change in Fasting Insulin Level | Baseline and after 12 weeks of intervention
  Fasting insulin will be measured to evaluate insulin levels at baseline and after 12 weeks of intervention
Change in HOMA-IR Index | Baseline and after 12 weeks of intervention
  HOMA-IR index will be calculated using fasting insulin and glucose levels to evaluate changes in insulin resistance.
Height in meters | Baseline only
  Height in meters will be measured using a stadiometer with participants standing without shoes, feet flat, and head positioned in the Frankfurt plane. The measurement will be recorded to the nearest 0.1 cm.
  The average height will be calculated for each group at baseline and used for descriptive comparison and used for BMI calculations.
Body fat percentage and lean body mass using bioelectrical impedance analysis (BIA) | Baseline and every 2 weeks until week 12
  Body composition, including body fat percentage and lean body mass, will be measured using a validated bioelectrical impedance analysis (BIA) device (InBody 120). Measurements will be conducted with participants fasting, at baseline and every 2 weeks during the 12-week intervention period.
  The mean and standard deviation for each variable will be calculated at each time point and compared between intervention groups over time.
Body Mass Index (BMI) in kg/m² | Baseline and every 2 weeks until week 12
  BMI will be calculated using the standard formula: weight (in kilograms) divided by the square of height (in meters) [kg/m²]. Weight and height will be measured using calibrated digital scales and stadiometers, respectively, with participants wearing light clothing and no shoes.
  The mean BMI will be calculated at each time point, and changes from baseline will be compared between intervention groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Aseel nutrition center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to privacy concerns and institutional policies. Data access is restricted to the research team to ensure confidentiality and compliance with ethical guidelines.